CLINICAL TRIAL: NCT04112069
Title: The Insulin-Only Bionic Pancreas Bridging Study- Pediatric Transitional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Clinical Study Director, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000853/JCHR
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Bionic pancreas; Closed loop; Insulin; Continuous glucose monitor
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Usual care (Active Comparator): Participants randomized to usual care first started the usual care arm (UC) managing their diabetes with continuous subcutaneous insulin infusion (pump therapy) for approximately 5 days. All subjects wore a Dexcom G5 continuous glucose monitor (CGM). If randomized to the usual care arm first, subjects crossed over to the bionic pancreas arm following a 2-day washout period.
  Interventions: Other: Usual Care
- iLet Bionic Pancreas with Humalog or Novolog (Experimental): Participants randomized to the iLet with humalog/novolog first started the insulin-only iLet arm using the insulin analog that they use for their usual care (either Humalog or Novolog) for approximately 5 days. All subjects wore a Dexcom G5 CGM. If randomized to the bionic pancreas arm first, subjects crossed over to the usual care arm following a 2-day washout period.
  Interventions: Device: iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog

INTERVENTIONS:
Device: iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog — iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog
  Arms: iLet Bionic Pancreas with Humalog or Novolog
Other: Usual Care — Usual care
  Arms: Usual care

SUMMARY:
The iLet is a closed-loop delivery system that can be used in insulin-only, bihormonal, or glucagon-only configurations. Previous studies have utilized a phone-based bionic pancreas. The iLet consists of a touchscreen-enabled, menu-driven user interface and an onboard microprocessor that provides a comprehensive and standalone platform, which allows the iLet to operate independently of smartphones or other devices and without the need for internet support during routine operation.

This is a multicenter study of pediatric participants with type 1 diabetes, who will manage their diabetes with the iLet bionic pancreas compared to usual care.

DETAILED DESCRIPTION:
20 pediatric participants from three clinical sites (Colorado, Nemours, and Stanford) will take part in the Pediatric Transitional Study Session to assess the efficacy, safety, and reliability of the insulin-only configuration of the bionic pancreas in regulating glycemia in pediatric subjects in a more supervised setting prior to beginning the true outpatient study. The Pediatric Transitional Study Session will consist of a multi-center, two-period, random-order, cross-over, pilot study in 20 pediatric participants 6-17 years old with T1D (~ 6 adolescent participants at Colorado 12-17 years old, ~ 6 pre-adolescent participants at Nemours 6-11 years old, and ~ 8 pediatrics subjects at Stanford 6-17 years old). Insulin therapy for each participant will be administered (i) in one period using the iLet in the insulin-only configuration with the iLet pigtail adapter and the iLet ready-to-fill insulin cartridge, the Contact Detach infusion set, the Dexcom G5 CGM, and the insulin analog that they use for their usual care (either Humalog or Novolog), and (ii) in the other period using the participant's own usual care (UC), where each participant will wear a Dexcom G5 CGM. Both experimental periods will be followed by round-the-clock, remote, telemetric monitoring for hyperglycemia (> 300 mg/dl for ≥ 90 minutes) and hypoglycemia (< 50 mg/dl for ≥ 15 minutes). The two experimental periods will each span 5 days, including 4 nights (e.g. Monday-Friday). A washout period of ~ 3 days in duration will separate the two experimental periods of the Pediatric Transitional Study Session.

Both study periods will be conducted in the same clinically supervised setting during each of the 5 days and at home under parental supervision or other overnight companion who is available to serve as an emergency contact during each of the 4 nights. Parents/guardians must be present (i.e. in the house or building) while the participant is home and sleeping and will serve as the contact person for overnight alerts. During the daytime in the Pediatric Transitional Study Session, participants of each cohort will be with the clinical study staff at each of the three clinical sites and will engage in common activities such that meals and activities can be well-characterized and supervised. For further quantification of stress due to exercise, activity monitors will be worn by all of the participants in both periods of the study. In terms of physical activity, diet, and remote monitoring for hypo- and hyperglycemia, parity will be maintained between both study periods.

All 20 pediatric participants in the Pediatric Transitional Study Session will use insulin pump therapy for their usual diabetes management. The Dexcom G5 CGM will serve as the input CGM to the iLet for all 20 pediatric participants. The cohort of 6 adolescent participants at Colorado and 6 pre-adolescent participants at Nemours, and 8 participants at Stanford might overlap or might not overlap in time.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year and using insulin for at least 1 year
2. Diabetes managed using an insulin pump for ≥ 3 months
3. Age 6-17 years
4. HbA1c level <11.0%

   • A point of care or local lab measurement is used to assess eligibility for screening.
5. At least 3 SMBG meter tests daily on average or use of a CGM and 2 or more SMBG meter tests daily on average by history
6. For females, not currently known to be pregnant

   • If female, sexually active, and at risk for pregnancy, must agree to use a highly effective form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all women who are post-menarche and pre-menopause who are not surgically sterile. Participants who become pregnant will be discontinued from the study.
7. An understanding of and willingness to follow the protocol and sign the informed consent and assent where applicable

Exclusion Criteria:

-The presence of any of the following is an exclusion for the study:

1. Unable to provide informed consent (e.g. impaired cognition or judgment)
2. Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the BP, impaired memory)
3. Unable to speak and read English
4. Currently using for the first time a real-time CGM for < 1 month (Individuals who have been using CGM for 1 or more months are eligible)
5. Current use of non-FDA approved closed-loop or hybrid closed-loop insulin delivery system
6. Current use of insulin glulisine (Apidra) as part of usual diabetes home regimen
7. Current off-label use of faster-acting insulin aspart (Fiasp) in CSII therapy as part of usual diabetes home regimen
8. Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the participant
9. Pregnant (positive urine HCG), breast feeding, plan to become pregnant in the next 12 months, or sexually active and at risk for pregnancy without use of contraception
10. Current alcohol abuse (intake averaging >4 drinks daily in last 30 days) or other substance abuse (use within the last 3 months of controlled substances other than marijuana without a prescription)
11. Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
12. Stage 4 renal failure (eGFR <30) or Stage 5 renal failure on dialysis (hemodialysis or peritoneal dialysis)
13. History of cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma, or history of complete pancreatectomy
14. Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. exercise of intensity up to 6 METS) despite medical management, or within the last 12 months before screening a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
15. Abnormal EKG consistent with increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, proximal LAD critical stenosis (Wellen's sign), or prolonged QT interval (> 440 ms). Other EKG findings, including stable Q waves, are not grounds for exclusion as long as the participant is not excluded according to other criteria. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.

    • EKG is only required for participants ≥50 years old or with diabetes duration ≥20 years
16. For participants < 50 years of age and < 20 years since diagnosis: History of prolonged QT interval, malignant arrhythmia, or congenital heart disease
17. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV
18. History of TIA or stroke in the last 12 months
19. Recent history of diabetic ketoacidosis (DKA) or severe hypoglycemia in the last 6 months. Severe hypoglycemia is defined as an event that required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma.
20. History of more than 1 episode of DKA requiring hospitalization in the last 2 years
21. History of more than 1 episode of severe hypoglycemia in the last year.
22. Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
23. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
24. Unable or unwilling to completely avoid acetaminophen for duration of study
25. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
26. History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
27. Current or planned use of SGLT2 inhibitors (prior use more than 3 months prior to enrollment is acceptable; SGLT2 inhibitors should not be initiated during the trial)
28. If using GLP1, pramlintide, or metformin must be on a stable dose for 3 months prior to enrollment (these agents should not be initiated during the trial)
29. Required use of 2 or more steroid bursts in the 6 months prior to the trial
30. History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
31. Any factors that, in the opinion of the site principal investigator or clinical protocol chair, would interfere with the safe completion of the study, including medical conditions that may require hospitalization during the trial

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Nemours Children's Specialty Care, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be published as online supplemental material to the main paper describing the results, as we have done for all of our previous bionic pancreas studies.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 pediatric participants
Pre-assignment Details: two-period, random-order, cross-over design. The two experimental periods each spanned5 days, including 4 nights (e.g. Monday-Friday). A washout period of ~ 3 days in duration separatedthe two experimental periods of the Pediatric Transitional Study Session.
Groups:
- Usual Care, Then iLet Bionic Pancreas With Humalog or Novolog: Usual Care first, then iLet Bionic Pancreas
  Participants randomized to usual care first started the usual care arm (UC) managing their diabetes with continuous subcutaneous insulin infusion (pump therapy) for approximately 5 days. If randomized to the usual care arm first, subjects switched to the bionic pancreas arm following a 2-day washout period.
- iLet Bionic Pancreas With Humalog or Novolog, Then Usual Care: iLet Bionic Pancreas first, then Usual Care
  Participants randomized to the iLet with humalog/novolog first started the insulin-only iLet arm using the insulin analog that they use for their usual care (either Humalog or Novolog) for approximately 5 days. If randomized to the bionic pancreas arm first, subjects switched to the usual care arm following a 2-day washout period.
  iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog: iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog
Period: Overall Study
Arm/Group | Usual Care, Then iLet Bionic Pancreas With Humalog or Novolog | iLet Bionic Pancreas With Humalog or Novolog, Then Usual Care
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: A two-period, random-order, cross-over design in 20 pediatric participants 7-17 years old with T1D
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (3)
Age, Customized [Number; unit: participants]
  age 14-17 years | 7
  age 10-15 years | 7
  age 7-11 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 13
  Hispanic or Latino | 3
  Asian | 3
  Native Hawaiian/Other Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean CGM Glucose
Description: Mean of all CGM data obtained with the Dexcom G5 through days 2-5 of the study
Time Frame: Days 2-5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
mg/dl | 159 (27) | 163 (15)

2. Primary Outcome: Percentage of Time With CGM Glucose Values <54 mg/dl
Time Frame: Days 2-5
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
percentage of time | 0.1 [0.0 to 0.4] | 0.4 [0.1 to 0.9]

3. Other Pre Specified Outcome: Percentage of Time Where CGM Glucose is Less Than 70 mg/dL
Time Frame: Day 2-5
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
percentage of time | 2.1 [0.7 to 5.1] | 1.7 [1.2 to 2.8]

4. Other Pre Specified Outcome: Percentage of Time in the Glucose Target Range of 70-180 mg/dl
Time Frame: Days 2-5
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
percentage of time | 65 (15) | 65 (10)

5. Other Pre Specified Outcome: Percentage of Time Where CGM Glucose is Greater Than 250 mg/dL
Time Frame: Day 2-5
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
percentage of time | 9 [3 to 12] | 9 [5 to 13]

6. Other Pre Specified Outcome: Percentage of Time Where CGM Glucose is Less Than 60 mg/dL
Time Frame: Day 2-5
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
percentage of time | 0.5 [0.3 to 1.4] | 0.6 [0.4 to 1.2]

7. Other Pre Specified Outcome: Number of Episodes of Severe Hypoglycemia
Description: Pre-specified to report the total number of episodes summed across all participants
Time Frame: Day 1-5
Measure: Number; unit: number of episodes
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
number of episodes | 3 | 6

8. Other Pre Specified Outcome: Number of Episodes of Diabetic Ketoacidosis (DKA)
Description: pre-specified to report the total number of episodes summed across all participants
Time Frame: Day 1-5
Measure: Number; unit: number of episodes
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
Number analyzed (Participants) | 20 | 20
number of episodes | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 months for the RCT (Randomized control trial)
Arm/Group | Usual Care | iLet Bionic Pancreas With Humalog or Novolog
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=20) | iLet Bionic Pancreas With Humalog or Novolog (N=20)
Hyperglycemia (Endocrine disorders) | 0 | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04112069/Prot_SAP_001.pdf